CLINICAL TRIAL: NCT00763750
Title: BrUOG-Brain-223-A Phase II Study of PPX (CT-2103), Temozolomide, and Concurrent Radiation for Newly Diagnosed Brain Tumors (CTI # CT2103) Principal Investigator: Howard Safran, M.D.
Brief Title: PPX, Temozolomide, and Concurrent Radiation for Newly Diagnosed Brain Tumors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: howard safran (Other)
Collaborators: Rhode Island Hospital (Other); MaineHealth (Other)
Responsible Party: Sponsor-Investigator, howard safran, Principle Investigator, Brown University
Organization: Brown University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BrUOG-Brain-223
Record Dates: First submitted 2008-09-30; First posted 2008-10-01 (Estimated); Results first posted 2013-12-16 (Estimated); Last update posted 2020-02-17 (Actual); Status verified 2020-02

CONDITIONS: Brain Tumor
Keywords: glioblastoma multiforme or anaplastic glioma
MeSH Terms: conditions — Brain Neoplasms; Glioblastoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- PPX +TMZ+XRT (Experimental): XRT 60Gy at 2 GY/fractions x 30 fractions TMZ 75mg/m2/day PPX 40mg/m2/week x 6 weeks Days 1,8,15,22,22,29,36
  Interventions: Drug: PPX +TMZ+XRT

INTERVENTIONS:
Drug: PPX +TMZ+XRT — PPX 50 mg/m2/week x 6 weeks (Days #1, 8, 15, 22, 29, 36) XRT: 60 Gy at 2 Gy/fraction x 30 fractions Temozolomide 75 mg/m2/day: Day #1 of XRT until completion (including weekends and holidays)
  Other Names: PPX TMZ

SUMMARY:
The purpose of this study is to determine the antitumor activity of PPX in combination with temozolomide and radiation for patients with newly diagnosed brain tumors.

DETAILED DESCRIPTION:
To evaluate the safety/tolerability and potential antitumor activity of PPX in combination with temozolomide and radiation for patients with newly diagnosed brain tumors.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histopathologically confirmed, newly diagnosed, glioblastoma multiforme or anaplastic glioma (anaplastic astrocytoma [AA], anaplastic oligodendroglioma, and anaplastic oligoastrocytoma) and have not had a complete surgical resection.
* Patients must be 18 years of age or older.
* Patients must have a Zubrod performance status 0-2.
* Patients must not be on enzyme-inducing anti-epileptic drugs (EIAED). Patients may be on non-enzyme inducing anti-epileptic drugs (NEIAED) or may not be taking any anti-epileptic drugs.
* Patients must not have received prior chemotherapy, radiation or any experimental therapy for their glioblastoma.
* Patients may not be breast-feeding a child.
* Female patients must either be not of child bearing potential or have a negative pregnancy test within 14 days of starting study treatment. Patients are considered not of child bearing potential if they are surgically sterile (they have undergone a hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) or they are postmenopausal. Pregnant or lactating females are not eligible. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
* Female patients must be using an acceptable method of contraception (oral contraceptives, barrier methods, approved contraceptive implant, long-term injectable contraception, intrauterine device or tubal ligation) OR female patients must be at least 1-year post-menopausal or surgically sterile during their participation in this study (from the time they sign the consent form) to prevent pregnancy. Male patients must be surgically sterile or using an acceptable method of contraception during their participation in this study (from the time they sign the consent form) to prevent pregnancy in a partner
* Patients must have no concurrent malignancy except curatively treated basal or squamous cell carcinoma of the skin or carcinoma in situ of the cervix or breast. Patients with prior malignancies must be disease-free for ≥ 2 years.
* Patients must have normal organ and marrow function as defined below:

  * Absolute neutrophil count > 1,500/ul
  * Platelets > 100,000/ul
  * Hemoglobin > 8 gm/dL
  * Total bilirubin < 1.5 x ULN
  * Creatinine < 1.5 x ULN
* Patient must have the capacity to understand and the willingness to sign a written informed consent document.
* Patient must be able to tolerate MRIs. CT scans can NOT be substituted for MRI in this study.

Exclusion Criteria:

* Recurrent malignant gliomas.
* Tumor foci detected below the tentorium or beyond the cranial vault.
* Allergy to gadolinium or contraindication to MRI scan.
* Patients who have received any form of brachytherapy or radiosurgery for their glioblastoma prior to start of standard radiation.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to PPX.
* Uncontrolled intercurrent illness including, but not limited to, hypertension ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant women are excluded from this study. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with PPX, breastfeeding should be discontinued if the mother is treated with PPX.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2008-10; Primary Completion 2011-06 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Howard Safran, MD, Principal Investigator — BrUOG
Locations (1):
- Lifespan Hospitals, Providence, Rhode Island, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- PPX +TMZ+XRT: XRT 60Gy at 2 GY/fractions x 30 fractions TMZ 75mg/m2/day PPX 40mg/m2/week x 6 weeks Days 1,8,15,22,22,29,36
  PPX +TMZ+XRT : PPX 50 mg/m2/week x 6 weeks (Days #1, 8, 15, 22, 29, 36) XRT: 60 Gy at 2 Gy/fraction x 30 fractions Temozolomide 75 mg/m2/day: Day #1 of XRT until completion (including weekends and holidays)
Period: Overall Study
Arm/Group | PPX +TMZ+XRT
Started | 25
Completed | 25
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | PPX +TMZ+XRT
Number analyzed (Participants) | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 17
  >=65 years | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 56 (5.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 12
Region of Enrollment [Number; unit: participants]
  United States | 25

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Assessed for Toxicity According to CTC Version 3.0
Time Frame: Throughout the entire study until patient is removed from study an average of 6 weeks
Measure: Number; unit: participants
Arm/Group | PPX +TMZ+XRT
Number analyzed (Participants) | 25
participants | 25

ADVERSE EVENTS:
Time Frame: Time of signing consent to 30 days post last dose of drug (approximately 4 months)
Arm/Group | PPX +TMZ+XRT
Serious Adverse Events (participants affected / at risk) | 6/25
Other Adverse Events (participants affected / at risk) | 25/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PPX +TMZ+XRT (N=25)
PLT gr 4, ANC 4, HGB 3 F/U: ANC to gr3, HGB and PLT to gr 2 (Investigations) | 1 (1)
gr 4 PLT, ANC 3, HGB2 & FU: death (Investigations) | 1 (1)
Plt gr4, ANC4, weakness/failure to thrive gr 3 & FU:gr 4 Leuko, gr 3 HGB, Anorexia gr 3, death (Investigations) | 1 (1)
weakness (gr 3) (Investigations) | 1 (1)
seizure - no grade (Investigations) | 1 (1)
gr 3 dehydration, gr 3 weakness, gr 3 Anorexia (Investigations) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PPX +TMZ+XRT (N=25)
rash (Investigations) | 5 (5)
infection normal ANC (thrush included) (Investigations) | 8 (8)
fatigue (Investigations) | 7 (7)
seizure (Investigations) | 3 (3)
headache (Investigations) | 3 (3)
insomnia (Investigations) | 2 (2)
vomiting (Investigations) | 2 (2)
Nausea (Investigations) | 2 (2)
Alopecia (Investigations) | 4 (4)
constipation (Investigations) | 3 (3)
Glucose (Investigations) | 5 (5)
Albumin (Investigations) | 4 (4)
Lymphopenia (Investigations) | 14 (14)
PLT (Investigations) | 4 (4)
ANC (Investigations) | 4 (4)
WBC (Investigations) | 4 (4)
HGB (Investigations) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No